CLINICAL TRIAL: NCT06934200
Title: Omalizumab for the Treatment of Food Allergy in Patients With Elevated Total IgE Levels
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00467873
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Food Hypersensitivity
Keywords: omalizumab
MeSH Terms: conditions — Food Hypersensitivity | interventions — Omalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with omalizumab (Other): This is an open label study of omalizumab with no placebo. Participants who meet study inclusion criteria and are enrolled in the study will receive omalizumab. The dose of omalizumab will be based on participant's weight.
  Interventions: Drug: Omalizumab

INTERVENTIONS:
Drug: Omalizumab — omalizumab injections

SUMMARY:
In this project, the investigators would like to learn if 24 weeks (about 5 and a half months) of omalizumab injections, given every 2 weeks, will be safe and effective for food allergic people who have a total immunoglobulin E (IgE) above the current FDA approved dosing regimen enabling a person to increase tolerance to the food(s) that the person is allergic to.

The investigators would also like to learn if participants who demonstrate increased tolerance to food after 24 weeks of omalizumab, can introduce the food into the diet utilizing an additional 8 weeks (about 2 months) of twice weekly omalizumab injections.

ELIGIBILITY:
Inclusion Criteria:

* Age 1 to 55 years
* A positive prick skin test (PST) with a wheal ≥ 6 mm to at least one of the relevant foods (peanut, cashew, walnut, egg, milk, or wheat)
* Positive food-specific IgE (≥2.0 kilo units of allergen-specific IgE per liter (kUA/L)) to at least one of the study specific foods
* A weight / IgE level that would have excluded the participant from the OUTMATCH study based on the dosing table noted above
* Positive double-blind, placebo-controlled food challenge (DBPCFC) to one of the relevant foods at a cumulative dose of ≤144 mg (maximum tolerated dose ≤30 mg)

Exclusion Criteria:

* Clinically significant laboratory abnormalities at screening.
* Dose-limiting symptoms during the blinded food challenge to placebo during the screening DBPCFC.
* Poorly controlled or severe asthma/wheezing at screening
* History of severe anaphylaxis to participant-specific foods that will be used in this study, defined as neurological compromise or requiring intubation.
* Treatment with a burst of oral, intramuscular (IM), or intravenous (IV) steroids of more than two days for an indication other than asthma/wheezing within 30 days of screening.
* Currently receiving oral, IM, or IV corticosteroids, tricyclic antidepressants, or β-blockers.
* Past or current history of eosinophilic gastrointestinal disease within three years of screening.
* Past or current history of cancer, or currently being investigated for possible cancer.
* Past or current history of any food immunotherapy (e.g., oral immunotherapy (OIT), sublingual immunotherapy (SLIT), epicutaneous immunotherapy (EPIT) within 6 months of screening.
* Treatment with monoclonal antibody therapy, such as omalizumab, dupilumab, benralizumab, mepolizumab, reslizumab, tezepelumab, or other immunomodulatory therapy within 6 months of screening.
* Inability to discontinue antihistamines for minimum wash-out periods required for skin prick tests (SPTs) or oral food challenges (OFCs).
* Pregnant or breastfeeding, or intending to become pregnant during the study
* Evidence of clinically significant chronic disease.

Ages: 1 Year to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants without dose limiting symptoms | 24 weeks
  Consumption of a single dose of 600mg or more of food protein without dose-limiting symptoms during the week 24 Double-blind, Placebo-controlled, Food Challenge

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wood, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wood RA, Togias A, Sicherer SH, Shreffler WG, Kim EH, Jones SM, Leung DYM, Vickery BP, Bird JA, Spergel JM, Iqbal A, Olsson J, Ligueros-Saylan M, Uddin A, Calatroni A, Huckabee CM, Rogers NH, Yovetich N, Dantzer J, Mudd K, Wang J, Groetch M, Pyle D, Keet CA, Kulis M, Sindher SB, Long A, Scurlock AM, Lanser BJ, Lee T, Parrish C, Brown-Whitehorn T, Spergel AKR, Veri M, Hamrah SD, Brittain E, Poyser J, Wheatley LM, Chinthrajah RS. Omalizumab for the Treatment of Multiple Food Allergies. N Engl J Med. 2024 Mar 7;390(10):889-899. doi: 10.1056/NEJMoa2312382. Epub 2024 Feb 25. PMID 38407394